CLINICAL TRIAL: NCT04025567
Title: Phase II Study of Oral Vancomycin in Patients With Unresectable Fibrolamellar Hepatocellular Carcinoma (FLC)
Brief Title: Vancomycin in Patients With Unresectable Fibrolamellar Hepatocellular Carcinoma (FLC) Oral
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow/insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190125; 19-C-0125
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Hepatocellular Carcinoma; Hepatocellular Carcinoma
Keywords: Gut Bacteria; Anti-Tumor Effects; NKT cells
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1 (Experimental): Oral vancomycin
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: vancomycin — 1,500 mg total daily dose, on days 1-21 of every 28 days cycle.

SUMMARY:
Background:

Fibrolamellar Hepatocellular Carcinoma (FLC) is a rare liver cancer. It most often occurs in young people who have no history of liver disease. Unresectable FLC most often does not improve with surgery. Researchers think gut bacteria may affect liver cancer control. They want to see if a drug that controls a type of bacteria can help.

Objective:

To test if vancomycin is safe and tolerable for and can treat people with unresectable FLC.

Eligibility:

People ages 18 and older with FLC that isn t responsive to treatment

Design:

Participants will be screened with a medical history, physical exam, blood and urine tests, and CT or MRI scans. They will provide a tumor sample: If they do not have one, they will have a biopsy.

Participants will take vancomycin 3 times a day. They will take the drug by mouth. They will take the drug in 28-day cycles. They will take the drug daily for the first 3 weeks. They will not take the drug the last week.

Participants will keep a medication diary.

Participants will have blood and urine tests each cycle. They may provide stool samples.

Participants will have a biopsy before they start treatment. Then they will have one on day 1 of cycle 2.

Participants will have scans on day 1 of cycle 2. Then they will have scans about every 8 weeks.

Participants will continue treatment until their cancer gets worse or they can no longer tolerate the side effects.

Participants will have a follow-up visit about a month after they finish treatment. Then they will be followed every 6 months by phone or email.

DETAILED DESCRIPTION:
Background:

* Fibrolamellar hepatocellular carcinoma (FLC) is a rare liver cancer (0.5-9% of primary liver cancers), which affects younger age groups and is not associated with underlying liver disease or elevated serum alpha fetoprotein (AFP) levels.
* Surgery, either liver resection (LR) or liver transplantation (LT), is the only potentially curative treatment for FLC patients with resectable disease. Disease recurrence after complete resection is high (33-100%). In patients with unresectable disease, median survival is less than 12 months; with no patient expected to survive beyond 5 years.
* The role of systemic chemotherapy and radiotherapy is poorly defined, and has been reported to have only a modest or no therapeutic effect. To date no targeted therapy has been shown to be of any value in FLC.
* In mouse models, oral vancomycin alters gut commensal bacteria thereby inducing a liver-selective anti-tumor effect by increasing hepatic CXCR6+ NKT cells via increased CXCL16 expression of liver sinusoidal endothelial cells.

Objective:

-To evaluate the effect of oral vancomycin therapy on the relative CXCR6 gene expression levels in the liver in paired pre- and on-treatment biopsy samples from hepatic lesions in patients with unresectable FLC

Eligibility:

* Histologically confirmed FLC, not amenable to potentially curative resection, transplantation or ablation.
* Liver lesion measurable by RECIST criteria, accessible for biopsy.
* Age greater than or equal to 18 years
* ECOG performance status less than or equal to 2
* Acceptable renal and normal liver function.
* Willingness to undergo pre- and on-treatment biopsies of liver tumor.

Design:

* This is a phase II study of oral vancomycin in patients with unresectable FLC.
* Up to 14 patients will be treated with oral vancomycin 500 mg tid daily (1,500 mg total daily dose) from days 1 to 21, in a 28-day cycles. After completion of the first cycle, initiation of concurrent treatment will be allowed. Patients will receive oral vancomycin until off treatment criteria are met.
* Patients will be evaluated for toxicity every 4 weeks by CTCAE v5.0, and for response at the end of the first cycle and thereafter every 8 (+/-3) weeks by RECIST 1.1.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of FLC by the NCI Laboratory of Pathology.
* Patients must have disease that is not amenable to potentially curative resection, transplantation or ablation.
* Patients must be greater than or equal to 18 years of age. Children are excluded from this study because this study has two mandatory biopsies performed for research purposes only and we do not want to put children into additional risk of biopsies.
* Patients must have evaluable or measurable hepatic disease per RECIST 1.1
* Patients must have hepatic lesion accessible for biopsy and be willing to undergo pre- and post-treatment mandatory biopsies.
* ECOG performance status of less than or equal to 2
* Adequate renal function defined by:

  * Creatinine <1.5 x institution upper limit of normal (ULN)
  * Creatinine clearance (CrCl) greater than or equal to 50 mL/min/1.73 m2 by 24 hours urine collection or eGFR as estimated using the chronic kidney disease (CKD)-EPI equation for participant with creatinine levels > 1.5 X institutional ULN.
* Adequate hepatic function defined by:

  * Total bilirubin level with upper limit of normal less than or equal to 1 (SqrRoot) ULN,
  * AST level <5(SqrRoot) ULN, and
  * ALT level <5 (SqrRoot) ULN.
* Adequate hematological function defined by:

  --Absolute neutrophil count (ANC) greater than or equal to 1.5 (SqrRoot) 109/L.
* Subjects must be co-enrolled onto protocol 11C0112.
* Ability of subject or Legally Authorized Representative to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had standard-of-care anti-cancer therapy (e.g., chemotherapy,immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents) within 2 weeks of enrollment; or, therapy with investigational agents, large field radiotherapy, or major surgery within 4 weeks prior to enrollment.
* Patients who are currently receiving any other investigational agents for any indication.
* Patients who are actively receiving broad-spectrum antibiotics or have received such within 4 weeks prior to enrollment.
* Patients with history of recurrent C. diff colitis
* Patients who are on anti-coagulation or anti-platelet medication that cannot be interrupted prior to study-specified biopsies, including:

  * Aspirin that cannot be discontinued for 7 days prior to biopsy
  * Clopidogrel and ticagrelor that cannot be discontinued for 5 days prior to biopsy
  * Ticlopidine that cannot be discontinued for 10 days prior to biopsy
  * Prasugrel that cannot be discontinued for 7 days prior to biopsy
  * Dipyridamole that cannot be discontinued for at least 2 days prior to biopsy
  * Cilostazol that cannot be discontinued for at least 3 days prior to biopsy
  * Coumadin that cannot be discontinued for 7 days prior to biopsy
  * Low molecular weight heparin (LMWH) that cannot be discontinued >24 hours prior to biopsy and unfractionated heparin (UFH) that cannot be discontinued >4 hours prior to biopsy. NOTE: LMWH or UFH may be used to transition patients on and off the above anti-coagulants, if deemed appropriate by the treating physician.
  * Oral direct thrombin inhibitor (dabigatran) or direct Factor Xa inhibitor (rivaroxaban, apixaban, and edoxaban) that cannot be discontinued for 4 days prior to biopsy
* Any other uncontrolled intercurrent illness or medical condition that per PI discretion would limit compliance with study requirements.
* Pregnant women are excluded from this study because this study has two mandatory biopsies performed for research purposes only and biopsies can have abortifacient effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-12 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of oral vancomycin therapy in the relative CXCR6 gene expression levels in the liver | 4 weeks
  Change from baseline to 4 weeks after starting treatment in the relative CXCR6 gene expression level in the liver as determined by mRNA with Nanostring

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0125.html